CLINICAL TRIAL: NCT07109921
Title: Effect of a Structured Early Rehabilitation Program on Long-Term Functional Recovery, Quality of Life, and Survival in Patients With Severe Acute Pancreatitis: A 5-Year Randomized Controlled Trial
Brief Title: Early Rehabilitation for Severe Acute Pancreatitis (ERN-SAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Hospital of Wuhan, Affiliated Hospital of Jianghan University (Other)
Responsible Party: Principal Investigator, Qiandi Huang, Principal investigator, Sixth Hospital of Wuhan, Affiliated Hospital of Jianghan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WHSHIRB-K-2019015
Record Dates: First submitted 2025-07-30; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Severe Acute Pancreatitis Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Early Rehabilitation Nursing (ERN) Group (Experimental): In addition to usual care, patients received a protocolized, multidisciplinary rehabilitation program initiated within 48 hours of ICU admission. The program consisted of progressive, goal-directed mobilization, respiratory therapy, and psychological support, delivered 7 days a week by trained nurses and physical therapists.
  Interventions: Behavioral: Structured Early Rehabilitation Nursing Program
- Active Comparator: Usual Care Group (Active Comparator): Patients received standard ICU care for SAP, including hemodynamic monitoring, mechanical ventilation, fluid management, nutritional support, and pain control. Rehabilitation was not protocolized and was provided only at the discretion of the treating physician.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Structured Early Rehabilitation Nursing Program — A protocolized, phased program. Phase 1 (unconscious): passive range of motion and repositioning. Phase 2 (awake/stable): respiratory training (deep breathing, incentive spirometry), bed mobility (bridging, rolling), and progressive mobilization (sitting at edge of bed). Phase 3 (active): in-place stepping and supervised ambulation. Psychological support was provided throughout. Safety criteria were monitored continuously.
  Arms: Experimental: Early Rehabilitation Nursing (ERN) Group
Other: Usual Care — Standard ICU management for SAP as directed by the primary ICU team. Rehabilitation was discretionary, typically limited to passive range of motion exercises by bedside nurses if deemed necessary.
  Arms: Active Comparator: Usual Care Group

SUMMARY:
This prospective, randomized controlled trial investigates the efficacy of a structured early rehabilitation nursing (ERN) program compared to usual care in patients with severe acute pancreatitis (SAP). Four hundred patients admitted to the intensive care unit (ICU) were randomized to either receive the ERN intervention or usual care. The study aims to evaluate the effects of ERN on ICU and hospital length of stay, systemic inflammation, physical function, long-term quality of life, and one-year survival.

DETAILED DESCRIPTION:
Patients with severe acute pancreatitis (SAP) often experience prolonged immobilization in the ICU, leading to complications such as ICU-acquired weakness (ICU-AW), extended hospital stays, and poor long-term functional outcomes. While early rehabilitation is beneficial in general critical care, its application in SAP is not well-established. This study was designed to address this gap by evaluating a comprehensive, structured early rehabilitation nursing (ERN) program. The program includes progressive mobilization, respiratory therapy, and psychological support, initiated within 48 hours of ICU admission. The hypothesis is that the ERN program, compared to usual care, will attenuate systemic inflammation, accelerate physical recovery, reduce length of stay, and lead to superior long-term functional independence, quality of life, and 1-year survival in patients with SAP.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years.
2. A diagnosis of SAP according to the 2012 revised Atlanta classification.
3. Admission to the ICU within 72 hours of symptom onset.
4. An anticipated ICU stay of more than 48 hours.

Exclusion Criteria:

1. Pre-existing conditions precluding rehabilitation (e.g., severe neuromuscular disease, unstable spinal fractures).
2. Acute myocardial infarction or unstable cardiac arrhythmia.
3. Intracranial hypertension.
4. Active gastrointestinal bleeding.
5. Pregnancy.
6. Patient or family refusal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
ICU Length of Stay (LOS) | From ICU admission to ICU discharge (assessed up to 90 days)
  Defined as the time from ICU admission to discharge, measured in days.
Hospital Length of Stay (LOS) | From hospital admission to hospital discharge (assessed up to 90 days)
  Defined as the total time from hospital admission to discharge, measured in days.

SECONDARY OUTCOMES:
Change in C-reactive protein (CRP) level | Baseline, Day 7
  Serum levels of CRP, measured in mg/L, to assess systemic inflammation.
Change in Interleukin-6 (IL-6) level | Baseline, Day 7
  Serum levels of IL-6, measured in pg/mL, to assess systemic inflammation.
Muscle Strength | At ICU discharge (within 24 hours prior to transfer from ICU)
  Assessed using the Medical Research Council (MRC) sum score, which ranges from 0 (complete paralysis) to 60 (normal strength). A score <48 indicates ICU-acquired weakness.
Change in Functional Independence | Baseline (at ICU admission), at hospital discharge, and at 3, 6, and 12 months post-discharge
  Assessed using the Barthel Index for Activities of Daily Living (ADL). The score ranges from 0 to 100, where higher scores indicate greater independence.
Change in Quality of Life | Baseline (at ICU admission), at hospital discharge, and at 3, 6, and 12 months post-discharge
  Measured using the World Health Organization Quality of Life-BREF (WHOQOL-BREF) instrument, which assesses physical health, psychological health, social relationships, and environment domains. Domain scores are transformed to a 0-100 scale, where higher scores indicate better quality of life.
One-Year All-Cause Mortality | Up to 12 months
  Number of deaths from any cause within 12 months of randomization.
Incidence of ICU-Acquired Complications | During ICU stay
  Number of patients experiencing pre-specified complications, including pressure ulcers, ventilator-associated pneumonia, and deep vein thrombosis.
Patient and/or Family Satisfaction | At hospital discharge (within 24 hours prior to discharge)
  Assessed using a validated 5-point Likert scale at discharge. The scale measures satisfaction with nursing care, ranging from 1 (very dissatisfied) to 5 (very satisfied). Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Hospital of Wuhan, Affiliated Hospital of Jianghan University, Wuhan, Hubei, China